CLINICAL TRIAL: NCT03088865
Title: Evaluation of an Internal Hospital Practice: The Effect of Altered Sampling Protocol on Blood Culture Contamination Rates: An Open, Randomized, Prospective Study
Brief Title: Evaluation of an Internal Hospital Practice: The Effect of Altered Test Tubes Sampling Order on Blood Culture Contamination Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0017-17-HMO
Record Dates: First submitted 2017-03-09; First posted 2017-03-23 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-02

CONDITIONS: Septicemia
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial Specimen Diversion (Experimental): Aspirating first blood volume into a regular blood collection tube
  Interventions: Diagnostic Test: aspirating first blood volume into a regular blood collection tube
- Standard practice (Active Comparator): Aspirating first blood into blood culture bottles (Standard practice)
  Interventions: Diagnostic Test: aspirating first blood volume into a regular blood collection tube

INTERVENTIONS:
Diagnostic Test: aspirating first blood volume into a regular blood collection tube — order of blood drawing

SUMMARY:
Implementation of the initial specimen diversion technique, in which the first milliliter of the venipuncture sample is not injected into the culture bottle, led to a significant reduction in blood culture contamination rates. This technique is based on the assumption that the skin plug aspirated during venipuncture is a major source of contaminating bacteria. One such diversion method is aspirating the first blood volume into a blood collection tube. It has, however, been suggested that regular blood collection tubes carry contaminants from the tube's stopper into the blood cultures drawn afterwards, thereby increasing contamination rates. The aim of this trial is to examine the effect of aspirating the first blood volume into a regular blood collection tube on blood culture contamination rate.

ELIGIBILITY:
Inclusion Criteria:

* Adults evaluated in the emergency room or as inpatients for suspected sepsis or having sepsis and from whom the treating physician plans to take, in the same venous puncture, blood cultures and additional blood tests (blood count and/or blood chemistry).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Blood culture contamination rate | 7 days
  A blood culture contamination is defined as growth in a single set of coagulase-negative Staphylococcus, Micrococcus, Viridans group Streptococcus, Propionibacterium acne, Corynebacterium sp (diphtheroids) or Bacillus sp.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Lalezari A, Cohen MJ, Svinik O, Tel-Zur O, Sinvani S, Al-Dayem YA, Block C, Moses AE, Oster Y, Salameh S, Strahilevitz J. A simplified blood culture sampling protocol for reducing contamination and costs: a randomized controlled trial. Clin Microbiol Infect. 2020 Apr;26(4):470-474. doi: 10.1016/j.cmi.2019.09.005. Epub 2019 Sep 17. PMID 31539635